CLINICAL TRIAL: NCT01519739
Title: Clinical Evaluation of Mediguide System in CRT Implants
Brief Title: Clinical Evaluation of Mediguide System in Cardiac Resynchronization Therapy (CRT) Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-11-043-EU-MG
Record Dates: First submitted 2012-01-18; First posted 2012-01-27 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MediGuide Arm (Experimental)
  Interventions: Device: MediGuide™

INTERVENTIONS:
Device: MediGuide™ — MediGuide™ system will be used to guide CRT implants

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the MediGuide™ system during CRT implants.

ELIGIBILITY:
Inclusion Criteria:

* Meet clinical indication for implantation of an SJM CRT system according to the current European Society of Cardiology (ESC) Guidelines for cardiac and resynchronization therapy
* Receiving a new implant or undergoing an upgrade from an existing ICD or pacemaker implant with no prior LV lead placement
* Ability to provide informed consent for study participation and are willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

* Currently participating in any other clinical study
* Have prosthetic valves
* Are pregnant or planning pregnancy in the next 1 month
* Are less than 18 years of age
* Have ventricular tachyarrhythmias resulting from transient or correctable factors such as drug toxicity, electrolyte imbalance, or acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The performance of the MediGuide™ system during CRT implant | 1 month post CRT implant
  Performance will be assessed in terms occurence of adverse events, easy of use and potential benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Herzzentrum Leipzig GmbH

REFERENCES:
- [Derived] Richter S, Doring M, Gaspar T, John S, Rolf S, Sommer P, Hindricks G, Piorkowski C. Cardiac resynchronization therapy device implantation using a new sensor-based navigation system: results from the first human use study. Circ Arrhythm Electrophysiol. 2013 Oct;6(5):917-23. doi: 10.1161/CIRCEP.113.000066. Epub 2013 Sep 3. PMID 24002003
- See also: Published paper (Circ Arrhythm Electrophysiol, 2013) for a feasibility study — http://www.ncbi.nlm.nih.gov/pubmed/24002003